CLINICAL TRIAL: NCT00532792
Title: A Randomized, Observer-Blind, Placebo-Controlled Study to Assess the Safety and Immunogenicity of Intramuscular Inactivated Influenza A/H5N1 Vaccine Administered With and Without an Adjuvant Patch in Healthy Adults
Brief Title: A/H5N1 Dose Ranging Study With Adjuvant Patch
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intercell USA, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLA101; HHSSO100200700031C
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-01

CONDITIONS: Pandemic Influenza
Keywords: Avian; Pandemic; Influenza; A/H5N1
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- Group 1 (Experimental)
  Interventions: Biological: A/H5N1
- Group 2 (Experimental)
  Interventions: Biological: A/H5N1
- Group 3 (Experimental)
  Interventions: Biological: A/H5N1
- Group 4 (Experimental)
  Interventions: Biological: A/H5N1
- Group 5 (Experimental)
  Interventions: Biological: A/H5N1
- Group 6 (Experimental)
  Interventions: Biological: A/H5N1
- Group 7 (Experimental)
  Interventions: Biological: A/H5N1
- Group 8 (Experimental)
  Interventions: Biological: A/H5N1
- Group 9 (Experimental)
  Interventions: Biological: A/H5N1
- Group 10 (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: A/H5N1 — Low dose A/H5N1 (0.5mL); Route IM - Day 0 and Day 21; No LT Patch Day 0 or Day 21
  Arms: Group 1
Biological: A/H5N1 — Low dose A/H5N1 (0.5mL); Route IM - Day 0 and Day 21; no LT patch on Day 0; LT Patch on Day 21
  Arms: Group 2
Biological: A/H5N1 — Low dose A/H5N1 (0.5mL); Route IM - Day 0 and Day 21; LT patch on Day 0 and Day 21
  Arms: Group 3
Biological: A/H5N1 — Medium dose A/H5N1 (0.5mL); Route IM - Day 0 and Day 21; no LT patch on Day 0 or Day 21
  Arms: Group 4
Biological: A/H5N1 — Medium dose A/H5N1 (0.5mL); Route IM - Day 0 and Day 21; no LT patch on Day 0; LT Patch on Day 21
  Arms: Group 5
Biological: A/H5N1 — Medium dose A/H5N1 (0.5mL); Route IM - Day 0 and Day 21; LT patch on Day 0 and Day 21
  Arms: Group 6
Biological: A/H5N1 — High dose A/H5N1 (0.5mL); Route IM - Day 0 and Day 21; no LT patch on Day 0 or Day 21
  Arms: Group 7
Biological: A/H5N1 — High dose A/H5N1 (0.5mL); Route IM - Day 0 and Day 21; no LT patch on Day 0; LT Patch on Day 21
  Arms: Group 8
Biological: A/H5N1 — High dose A/H5N1 (0.5mL); Route IM - Day 0 and Day 21; LT patch on Day 0 and Day 21
  Arms: Group 9
Biological: Placebo — Placebo (0.5ml); Route IM - Day 0 and Day 21; no LT patch on Day 0 or Day 21
  Arms: Group 10

SUMMARY:
This is a Phase 1/2, randomized, observer-blind, placebo-controlled clinical trial. A maximum of 500 eligible subjects in 10 groups will be enrolled, randomized and vaccinated in this study. Subjects will receive an intramuscular injection of either the influenza A/H5N1 (low, medium or high dose) or placebo on Day 0 and Day 21 with or without a patch. This study will be performed in two parts.

In Part 1, an initial safety evaluation will be performed in 100 randomized subjects. A Safety Review Committee (SRC)will review all safety data, including laboratory values, through the Day 7 visit, and compare those data against Stopping Criteria. If the treatments are considered safe, Part 2 of the study will be initiated and a second vaccination will be administered to subjects in Part 1 on Day 21.

In Part 2, the remaining 400 subjects will be randomized, treated, and will follow the same visit structure and protocol-defined requirements as subjects in Part 1, without the additional laboratory safety measurements. An SRC review will also be performed of all safety data through the Day 28 visit for subjects participating in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females 18-49 years of age (inclusive)
* Signed Informed Consent
* Women who are not post-menopausal or surgically sterile must have a negative serum or urine pregnancy test at screening and within 24 hours of each vaccination with understanding (through Informed Consent process) to not become pregnant and to employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: abstinence, hormonal contraceptives (oral, injectable, implant, patch, ring), double-barrier contraceptives (condom or diaphragm, with spermicide), and IUD

Exclusion Criteria:

* Laboratory abnormalities [as determined by the Toxicity Grading Scale (grade 1 4)] at laboratory screening
* Abnormalities at physical examination [as determined by the Toxicity Grading Scale (grade 1-4)]
* Known allergies to any component of the vaccine
* Known egg protein allergy
* Known allergies to adhesives
* Known disturbance of coagulation
* Participated in research involving investigational product within 45 days before planned date of first vaccination
* Donated or received blood or blood products such as plasma within the past 45 days
* Received any licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to planned date of first vaccination
* Ever received investigational enterotoxigenic E. coli, LT, or LT (R192G) or NasalFlu, Berna Biotech, Ltd
* Ever received cholera toxin or vaccine (e.g. Orochol™, Dukoral™)
* History of travelers' diarrhea in the last two years
* History of abdominal surgery (excluding C-section, hysterectomy, cosmetic surgery, liposuction, appendectomy, cholecystectomy, ventral hernia repair, and other surgeries not pertaining to gastrointestinal problems) or history of, or recent acute gastrointestinal illness
* Previous vaccination with a pandemic candidate vaccine or previous proven contact with A/H5N1 wild type virus (contact with an individual with laboratory-confirmed A/H5N1 infection or contact with an animal which died as a result of A/H5N1 infection)
* Recent or regular use of oral, topical or injected steroid medications within 45 days prior to first vaccination
* Use of immunosuppressive systemic steroid medications including inhaled steroids within three months prior to first vaccination
* Comorbid conditions or treatments that are immunosuppressive, including cancer, diabetes, end-stage renal disease, as determined by the Investigator
* Positive serology for HIV-1, HIV-2, HBsAg, or HCV
* History of severe atopy
* Medical history of acute or chronic skin disease at vaccination area(s)
* Active skin allergy
* Signs of acute skin infection, sunburn or skin abnormalities at the vaccination area(s) including fungal infections, severe acne, or active contact dermatitis, or a history of keloid formation
* Hirsute (significant amount of hair) at vaccination area(s)
* Artificial tanning (UV radiation) over the duration of the study including the screening period
* Visible tattoos or marks (tattoos/scars) at the vaccination area(s) that would prevent appropriate dermatologic monitoring of the vaccination site(s)
* Fever greater than or equal to 38.0°C (100.4°F) at the time of planned vaccination
* Suspicion of or recent history of (within one year of planned vaccination) alcohol or substance abuse
* Women who are pregnant or breastfeeding
* Acute illness at screening or at baseline
* Ever had a serious reaction to prior influenza vaccination
* Developed a neurological disorder (such as Guillain Barré syndrome) in the six weeks following a previous influenza vaccination
* Medical history of achlorhydria
* Employee of the investigational site
* History of employment in bird or poultry industries or considerable exposure to birds (e.g. poultry or bird veterinarians, bird breeders, poultry butchers and/or cullers, etc.)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 501 (Actual)
Dates: Start 2007-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety of Intramuscular A/H5N1 with and without the LT adjuvant patch | 6 months

SECONDARY OUTCOMES:
Demonstration of adjuvant effect and evaluation of immunogenicity | Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Philip Leese, MD, Principal Investigator — Quintiles Phase One Services
Locations (5):
- United States (5):
  - Solano Clinical Research, Vallejo, California
  - Miami Research Associates, Miami, Florida
  - Quintiles Phase One Services, Kansas City, Kansas
  - Jean Brown Research, Salt Lake City, Utah
  - Northwest Kinetics, Tacoma, Washington